CLINICAL TRIAL: NCT07288827
Title: A Multi-center Study Examining Bronchial Hyperresponsiveness in Primary Ciliary Dyskinesia
Brief Title: Examining Bronchial Hyperresponsiveness in Primary Ciliary Dyskinesia
Acronym: BHR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Evans Machogu, Professor of Clinical Pediatrics, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16122
Record Dates: First submitted 2025-11-20; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Primary Ciliary Dyskinesia; Healthy
Keywords: Primary Ciliary Dyskinesia; bronchial hyperresponsiveness
MeSH Terms: conditions — Ciliary Motility Disorders; Bronchial Hyperreactivity | interventions — Phlebotomy; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Subjects with Primary Ciliary Dyskinesia and Healthy subjects (controls)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects with Primary Ciliary Dyskinesia (Experimental): Subjects will come to Riley Hospital for Children for at least two visits with the opportunity for a third visit. Each visit should take between 2 and 2.5 hours. During the visits, subjects will complete multiple breathing tests, inhale certain medications, complete a family history questionnaire, have skin allergy testing, and do a blood draw.
  Interventions: Procedure: Lung Function Testing; Procedure: Phlebotomy; Procedure: Allergy skin prick testing; Procedure: Methacholine Challenge
- Healthy Subjects (Experimental): Subjects will come to Riley Hospital for Children for at least two visits with the opportunity for a third visit. Each visit should take between 2 and 2.5 hours. During the visits, subjects will complete multiple breathing tests, inhale certain medications, complete a family history questionnaire, have skin allergy testing, and do a blood draw.
  Interventions: Procedure: Lung Function Testing; Procedure: Phlebotomy; Procedure: Allergy skin prick testing; Procedure: Methacholine Challenge

INTERVENTIONS:
Procedure: Lung Function Testing — will include baseline spirometry (pre- and post- max bronchodilator). All testing will be done according to American Thoracic Society/European Respiratory Society guidelines. Participants will be asked to refrain from taking any asthma medications, including inhaled corticosteroids, short- and long-acting bronchodilators, leukotriene receptor antagonists, and long-acting muscarinic antagonists, for 24 hours prior to any spirometry. This activity will take place at a clinical research center at the respective participating institution.
  Other Names: spirometry
Procedure: Phlebotomy — will be obtained at visit 2. Up to ten (10) ml of blood will be collected for measurement of serum biomarkers of atopy, based on whether participants prefer to receive an allergy skin prick test or have antigen-specific IgE levels tested. In the event a subject refuses phlebotomy, historical results up to one year old may be used in lieu of prospective results. Any remaining blood samples will be banked either for use in future studies or in the event that additional serum biomarkers are added to this study.
  Other Names: blood draw
Procedure: Allergy skin prick testing — may be completed at visit 2. Subjects will be instructed to withhold first-generation antihistamines for 3 days and second-generation antihistamines for 7 days prior to the test. If patients prefer to have serum antigen-specific IgE levels run with the required serum biomarkers of atopy, then skin prick testing will be omitted.
Procedure: Methacholine Challenge — If the subject does not demonstrate a bronchodilator response in FEV1 of 10% or greater, and does not have a historical MCT on file, MCT will be performed. Following inhalation of saline, methacholine (MCh) will be inhaled in quadrupling concentrations starting with 0.0625 mg/ml and continuing until the MCh concentration required for FEV1 to decrease by 20% from baseline (PD20) is achieved or a maximum MCh concentration of 16 mg/ml is inhaled.
  Other Names: MCT

SUMMARY:
The purpose of this study is to look at children with PCD and see if they have another condition called "bronchial hyperresponsiveness".

DETAILED DESCRIPTION:
The purpose of this study is to look at children with PCD and see if they have another condition called "bronchial hyperresponsiveness". This is when some of the air tubes ("bronchi") are very sensitive ("hyperresponsive") to certain things in the environment such as pollen, mold, pet dander, changes in temperature, and viruses. Children with PCD are often prescribed daily inhaled steroids to help make their air tubes less sensitive, but there are few research studies showing that children with PCD really need this medication.

In this study, the investigators will simulate the above triggers for sensitive air tubes with a medication called methacholine. Checking how fast children can breathe out after giving methacholine is sometimes done when doctors think a child may have asthma, a condition where the breathing tubes are very sensitive. By measuring the participant's breathing before and after giving this medication, the investigators will see whether their air tubes are sensitive, or "hyperresponsive". It is possible that methacholine could make the participants temporarily feel short of breath or start wheezing. To avoid this, the investigators will start by giving a small dose of methacholine and measuring the participants breathing, then give larger amounts of methacholine until the investigators see certain changes in the participants breathing or until the largest dose allowed is reached. If the participant starts to have symptoms such as shortness of breath, chest tightness, or wheezing, the investigators will give them a medicine called albuterol which immediately opens the air tubes and makes the symptoms go away. Any discomfort caused by the methacholine is temporary and there are no long-term effects associated with using it.

If the participants agree to participate in the study, they will come to Riley Hospital for Children for at least two visits with the opportunity for a third visit. Each visit should take between 2 and 2.5 hours. During the visits, they will complete multiple breathing tests, inhale certain medications, complete a family history questionnaire, have skin allergy testing, and do a blood draw.

The investigators will also collect information about the participants from your medical record, including demographic information, medical history, and disease history. If they have completed pulmonary function testing (testing that shows how well lungs are working) in the past, they may only be eligible for Visit 1.

For scheduling convenience, visits 1 and 2 may occur on the same day. The participants will be in this study up to one month if they participate in visits 1 and 2, and up to five months if they are eligible for visit 3.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PCD per standard diagnostic criteria4 and positive genetics
* Age greater than or equal to 6 years (no upper age limit)
* Any gender or race
* Able to perform pulmonary function testing (historical documentation of reversibility will be accepted)

Exclusion Criteria:

* history of current pneumothorax
* inability to perform pulmonary function testing

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Bronchial Hyperresponsiveness prevalence | From spirometry baseline measurement (Visit 2) to completion of post-max bronchodilator test (Visit 2) (<1hr)
  Examine how many subjects with PCD have bronchial hyperresponsiveness as evidenced by an increase in FEV1 of 10% or greater during pre- and post- max bronchodilator test.
Bronchial Hyperresponsiveness prevalence | From spirometry baseline measurement (Visit 3) to completion of methacholine challenge test (Visit 3) (<1hr)
  Examine how many subjects with PCD have bronchial hyperresponsiveness as evidenced by a decline in FEV1 by 20% from baseline during methacholine challenge test.
Bronchial Hyperresponsiveness prevalence | From spirometry baseline measurement (Visit 2) to completion of post-max bronchodilator test (Visit 2) (<1hr)
  Examine how many healthy subjects have bronchial hyperresponsiveness as evidenced by an increase in FEV1 of 10% or greater during pre- and post- max bronchodilator test.
Bronchial Hyperresponsiveness prevalence comparison | From first Visit 2 baseline measurement of first subject enrolled to either: last Visit 3 visit of PCD subject who may complete Visit 3; or last Visit 2 visit of PCD subject or Healthy subject, whichever comes latest in enrollment (up to five years)
  Compare the prevalence of bronchial hyperresponsiveness (examined in Outcome 1, Outcome 2) in PCD subjects to bronchial hyperresponsiveness in age- and gender-matched healthy controls.

SECONDARY OUTCOMES:
Data Collection of PCD genotype/phenotype | From first Visit 2 baseline measurement of first subject enrolled to either: last Visit 3 visit of PCD subject who may complete Visit 3; or last Visit 2 visit of PCD subject or Healthy subject, whichever comes latest in enrollment (up to five years)
  These data points will be a compilation of chronic rhinosinusitis, respiratory distress at birth, recurrent upper and lower airway infections, and/or fertility issues, serum biomarkers for atopy, and other clinical features and explore the relationship between PCD and bronchial hyperresponsiveness, which can manifest as coughing, wheezing, and/or chest tightness.
Analysis of the relationship between PCD and atopy | From first Visit 2 baseline measurement of first subject enrolled to either: last Visit 3 visit of PCD subject who may complete Visit 3; or last Visit 2 visit of PCD subject or Healthy subject, whichever comes latest in enrollment (up to five years)
  This will address whether bronchial hyperresponsiveness in PCD is due to an underlying predisposition similar to that seen in asthma and whether it could relate to some other mechanism such as antigen mucostasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States